CLINICAL TRIAL: NCT04869059
Title: Treatment of Verbal Retrieval Deficits in Mild Traumatic Brain Injury With High Definition Transcranial Direct Current Stimulation
Brief Title: Treating Mild Traumatic Brain Injury With High Definition Transcranial Direct Current Stimulation
Acronym: HDtDCS-TBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, John Hart, Jr., Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UTD-TDCSTBI-21-15; CDMRP-PT190081 (Other: CDMRP); W81XWH-20-1-0846 (Other Grant/Funding Number: DOD-CDMRP-USAMRDC)
Record Dates: First submitted 2021-02-10; First posted 2021-05-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; transcranial direct current stimulation; electroencephalography; cognition; veteran traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 treatment arms: (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 15 sessions to (2) sham tDCS following the same schedule.
  Additionally, after completing the initial active or sham treatment and 3-month follow-up testing sessions, selected participants will be invited back for newly assigned treatment conditions, 20 minutes over 15 sessions and will be and re-evaluated at 2- and 3-months follow-up testing sessions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, assessors, and technicians interacting with participants will be blind to assigned conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial direct current stimulation (Experimental): 20 minutes of 1 milliamp transcranial direct current stimulation to presupplementary motor area for 15 sessions
  Interventions: Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): 20 minutes of sham transcranial direct current stimulation to presupplementary motor area for 15 sessions
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. Stimulation will consist of 1 milliamp stimulation, with anodal stimulation delivered at electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, then remain at 1 milliamp of stimulation over 20 minutes, and finally ramping down at to 0 milliamps over 60 seconds.
  Other Names: tDCS; 1 milliamp tDCS; High definition tDCS; High definition transcranial direct current stimulator, Neuroelectrics Starstim tES, SN E20200930-10
  Arms: Transcranial direct current stimulation
Device: sham tDCS — Sham transcranial direct current stimulation will be delivered via a Neuroelectrics Starstim tES. The sham setup will consist of anodal electrode Fz (International 10/10 System for electroencephalography electrode placement) and electrodes F7, FP1, FP2, and F8 as returns. All electrodes are 1 cm diameter Ag/AgCl electrodes and make contact with the scalp via connective gel. Stimulation will linearly ramp up from 0 milliamps to 1 milliamp over 60 seconds, ramp down to 0 milliamps over 60 seconds and then be left off for 20 minutes.
  Arms: Sham transcranial direct current stimulation

SUMMARY:
The purpose of the study is to test whether low level electric stimulation, called transcranial Direct Current Stimulation (tDCS), on the part of the brain (i.e., presupplementary motor area) thought to aid in memory will improve verbal retrieval in military veteran participants with histories of traumatic brain injuries. The primary outcome measures are neuropsychological assessments of verbal retrieval, and the secondary measures are neuropsychological assessments of other cognitive abilities and electroencephalography (EEG) measures. Additionally, the study will examine the degree to which baseline assessments of cognition and concussion history predict responses to treatment over time, both on assessments administered within the intervention period and at follow-up.

DETAILED DESCRIPTION:
Using two treatment arms, the study will examine improvement of verbal retrieval and other cognitive deficits associated with remote traumatic brain injury by comparing (1) 1 milliamp transcranial direct current stimulation (tDCS) active treatment applied to presupplementary motor area for 20 minutes over 15 sessions to (2) sham tDCS following the same schedule. Additionally, after completing the initial active or sham treatment and 3-month follow-up testing sessions, selected participants will be invited back for newly assigned treatment conditions, 20 minutes over 15 sessions and will be and re-evaluated at 2- and 3-months follow-up testing sessions.

Veterans with histories of traumatic brain injuries and observed cognitive deficits will be randomly assigned to one of the two treatment arms (and re-assigned for the second round of intervention, as described above). Primary outcome verbal retrieval measures, secondary neuropsychological and electroencephalography (EEG) measures, and prescreening assessments for study concussion history and contraindications for treatment will be collected prior to being assigned to a treatment arm (i.e., baseline).

Primary outcome verbal retrieval measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected after treatment sessions 5, 10, and 15 and two times following treatment competition (i.e., 2-months and 3-months). For participants selected for the second round of intervention, primary outcome verbal memory measures and secondary neuropsychological and electroencephalography (EEG) measures will be collected again after treatment sessions 5, 10, and 15 and two times following competition of the second treatment (i.e., 2-months and 3-months).

ELIGIBILITY:
Inclusion Criteria: Participants are to be between the ages of 18-75, have previously served in the US armed services, and have had a traumatic brain injury that has led to a verbal retrieval deficit based on neuropsychological testing criteria. Traumatic brain injury must be in the mild to moderate range based on evaluation, including, the Ohio State TBI Identification Method (administered by our research group). You must be fluent in speaking and reading English.

Exclusion Criteria: Exclusion criteria include a history of a psychological or neurological disorder, including, dementia of any type, epilepsy or other seizure disorders, severe traumatic brain injury, post-traumatic stress disorder, brain tumor, present drug abuse, stroke, blood vessel abnormalities in the brain, Parkinson's disease, Huntington's disease, or multiple sclerosis. Additionally, exclusion criteria include inability to give informed consent; cranial implants or skull defects that affect tDCS administration; and use of medications that interact with or potentially interact with tDCS effects, including, anti-convulsants, amphetamines, L-dopa, carbamazepine, sulpiride, pergolide, lorazepam, rivastigmine, dextromethorphan, D-cycloserine, flunarizine, ropinirole, or citalopram.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Controlled Oral Word Association Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Control Word Association Test from baseline to 3-months. Metric: Number of Correct Items Generated
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Controlled Oral Word Association Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Control Word Association Test from baseline to 2-months. Metric: Number of Correct Items Generated
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
Treatment group differences in change from Baseline to 3-months Post-Treatment in Category Fluency | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Category Fluency from baseline to 3-months. Metric: Number of Correct Items Generated
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
Treatment group differences in change from Baseline to 2-months Post-Treatment in Category Fluency | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Category Fluency from baseline to 2-months. Metric: Number of Correct Items Generated
  Benton, L.A., Hamsher, K., & Sivan, A.B., (1994). Multilingual aphasia examination. Iowa City: AJA Associates.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Semantic Object Retrieval Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Semantic Object Retrieval Test from baseline to 3-months. Metric: Number of Correct Retrievals
  Kaplan, E., Goodglass, H., & Weintraub, S., (1983). Boston Naming Test (2nd ed.). Lea & Febiger: Philadelphia.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Semantic Object Retrieval Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Semantic Object Retrieval Test from baseline to 2-months. Metric: Number of Correct Retrievals
  Kaplan, E., Goodglass, H., & Weintraub, S., (1983). Boston Naming Test (2nd ed.). Lea & Febiger: Philadelphia.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Boston Naming Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Boston Naming Test from baseline to 3-months. Metric: Number of Correct Names Retrieved
  Kraut, M.A., Cherry, B., Pitcock, C.B., Anand, R., Li, J. Vestal, L., Henderson, V.W., and Hart, J. Jr. (2007). The Semantic Object Retrieval Test (SORT) in amnestic cognitive impairment. Cogn. Behav. Neurol. 20, 62- 67.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Boston Naming Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Boston Naming Test from baseline to 2-months. Metric: Number of Correct Names Retrieved
  Kraut, M.A., Cherry, B., Pitcock, C.B., Anand, R., Li, J. Vestal, L., Henderson, V.W., and Hart, J. Jr. (2007). The Semantic Object Retrieval Test (SORT) in amnestic cognitive impairment. Cogn. Behav. Neurol. 20, 62- 67.
Treatment group differences in change from Baseline to 3-months Post-Treatment on California Verbal Learning Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in California Verbal Learning Test from baseline to 3-months. Metric: Number of Correct Retrievals
  Delis DC, Kramer JH, Kaplan E, Ober BA. (2017). California verbal learning test (3rd Ed.). Pearson Publishing: San Antonio, TX.
Treatment group differences in change from Baseline to 2-months Post-Treatment on California Verbal Learning Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in California Verbal Learning Test from baseline to 2-months. Metric: Number of Correct Retrievals
  Delis DC, Kramer JH, Kaplan E, Ober BA. (2017). California verbal learning test (3rd Ed.). Pearson Publishing: San Antonio, TX.

SECONDARY OUTCOMES:
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Trail Making Test (Part A) | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part A) from baseline to 3-months. Metric: Time to Solution
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Trail Making Test (Part A) | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part A) from baseline to 2-months. Metric: Time to Solution
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Trail Making Test (Part B) | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part B) from baseline to 3-months. Metric: Time to Solution
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Trail Making Test (Part B) | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part B) from baseline to 2-months. Metric: Time to Solution
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Delis Kaplan Color Word Interference Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Delis Kaplan Color Word Interference Test from baseline to 3-months. Metric: Time to Name Items
  Delis, D.C., Kaplan, E., & Kramer, J.H., (2001). Delis-Kaplan Executive Function System. San Antonio, TX: The Psychological Corporation.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Delis Kaplan Color Word Interference Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Trail Making Test (Part B) from baseline to 2-months. Metric: Time to Name Items
  Reitan, R.M., (1958). Validity of the Trail Making Test as an indicator of organic brain damage. Percept. Motor Skill., 8, 271-276.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Digit Span Forward | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Digit Span Forward from baseline to 3-months. Metric: Memory Span
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Span Forward | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Digit Span Forward from baseline to 2-months. Metric: Memory Span
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Digit Span Backward | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Digit Span Backward from baseline to 3-months. Metric: Memory Span
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Span Backward | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Digit Span Backward from baseline to 2-months. Metric: Memory Span
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Rey-Osterrieth Complex Figure Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change in Rey-Osterrieth Complex Figure Test scores from baseline to 3-months. Metric: Score
  Rey, A. (1941). L'examen psychologique dans les cas d'encéphalopathie traumatique. (Les problems.). [The psychological examination in cases of traumatic encepholopathy. Problems.]. Archives de Psychologie, 28, 215- 285.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Rey-Osterrieth Complex Figure Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change in Rey-Osterrieth Complex Figure Test scores from baseline to 2-months. Metric: Score
  Rey, A. (1941). L'examen psychologique dans les cas d'encéphalopathie traumatique. (Les problems.). [The psychological examination in cases of traumatic encepholopathy. Problems.]. Archives de Psychologie, 28, 215- 285.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Digit Symbol Substitution Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Digit Symbol Substitution Test from baseline to 3-months. Metric: Number of Items
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Digit Symbol Substitution Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Digit Symbol Substitution Test from baseline to 2-months. Metric: Number of Items
  Wechsler, D., (2008). Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio, TX: NCS Pearson.
Treatment group differences in change from Baseline to 3-months Post-Treatment on the Grooved Pegboard Test | Outcome measures will be assessed as change over a period of 17 weeks: Change from baseline to 3-month Post-Treatment
  Evaluation of treatment group differences in change on the Grooved Pegboard Test from baseline to 3-months. Metric: Completion Time
  Matthews, C.G., and Klove, H. (1964). Instruction manual for the adult neuropsychology test. Madison. Wis: University of Wisconsin Medical School.
Treatment group differences in change from Baseline to 2-months Post-Treatment on the Grooved Pegboard Test | Outcome measures will be assessed as change over a period of 13 weeks: Change from baseline to 2-month Post-Treatment
  Evaluation of treatment group differences in change on the Grooved Pegboard Test from baseline to 2-months. Metric: Completion Time
  Matthews, C.G., and Klove, H. (1964). Instruction manual for the adult neuropsychology test. Madison. Wis: University of Wisconsin Medical School.

CONTACTS AND LOCATIONS:
Overall Officials: John Hart, MD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Dallas, Texas, United States